CLINICAL TRIAL: NCT00781963
Title: Implementing Sleep Interventions for Older Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 08-295
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Insomnia
Keywords: cognitive behavior therapy; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-I (Experimental): Manual-based cognitive behavioral therapy for insomnia (CBT-I) provided in 5 individual or group sessions by a non-clinician sleep coach.
  Interventions: Behavioral: Manual-based cognitive behavioral therapy for insomnia
- Control (Active Comparator): Non-directive sleep education provided in 5 group sessions by a health educator.
  Interventions: Behavioral: Non-directive sleep education

INTERVENTIONS:
Behavioral: Manual-based cognitive behavioral therapy for insomnia — Manual-based CBT-I provided in 5 individual or group sessions by a non-clinician sleep coach.
  Arms: CBT-I
Behavioral: Non-directive sleep education — Manual-based non-directive sleep education provided in 5 group sessions by a health educator.
  Arms: Control

SUMMARY:
Sleep problems are common among older people, and research suggests that insomnia has negative effects on health and quality of life in older adults. Prior research suggests that insomnia symptoms are even more common among veterans compared to the general population. In addition, people with sleep problems also often have depression and other problems that seem to decrease their quality of life. In this study, we tested two methods of providing behavioral sleep interventions for treating insomnia in older veterans. The long-term objective of this work was to identify ways to improve access to these types of behavioral sleep interventions for older veterans, in order to improve their well-being and quality of life. This project was conducted in outpatient clinics of the VA Greater Los Angeles Healthcare System. Community-dwelling older veterans (aged 60 years and older) with insomnia were identified by a postal survey. Enrolled veterans with insomnia (N=150 total, 50 per group) were randomized to one of three groups: Individual-Cognitive Behavioral Therapy for Insomnia (Individual-CBTI), Group-CBTI or a group-based Sleep Education Control Condition (Control). Measures of sleep, depression and quality of life were performed at baseline (enrollment in the study), after the treatment was completed, and at 6-months and 12-months follow-up after randomization. Main outcome measures included sleep/wake patterns (sleep questionnaires, sleep diary and wrist actigraphy, which is an objective estimate of sleep and wakefulness). We hypothesized that the intervention would improve sleep at six months follow-up. We also expected that these improvements would be maintained at 12-months follow-up.

DETAILED DESCRIPTION:
Sleep disturbance is common among older people due to age-related changes in sleep, in addition to health conditions, psychosocial issues, medication effects and a variety of other factors that impact sleep. The evidence that insomnia has negative effects on health and quality of life in older adults is convincing. Prior research has demonstrated that insomnia symptoms are even more common among veterans compared to the general population. Our own work has demonstrated that sleep problems are associated with depressive symptoms and other impairments in quality of life in older people, and that nonpharmacological and behavioral interventions can improve sleep in a variety of settings.

Objectives: We tested two methods of providing behavioral sleep interventions for treating insomnia in older veterans. The long-term objective of this work was to identify ways to improve access to behavioral sleep interventions for older veterans, in order to improve their well-being and quality of life.

Methods: This project was conducted in outpatient clinics of the VA Greater Los Angeles Healthcare System. Community-dwelling older veterans (aged 60 years and older) with insomnia were identified by a postal survey. Enrolled veterans with insomnia (N=150, 50 per group) were randomized to one of three groups:Individual Cognitive Behavioral Therapy for Insomnia (Individual-CBTI), Group-CBTI, or group-based Sleep Education Control Condition (Control). The intervention involved a manual-based behavioral sleep intervention provided by a non-clinician sleep coach. Baseline data included subjective and objective measures of sleep, and structured assessments of depression and quality of life. Post-treatment assessments was performed after completion of the 6-week intervention, and follow-up assessments were performed at 6-months and 12-months after randomization. Main outcome measures were: sleep measures obtained from sleep diaries (i.e., sleep onset latency, wake after sleep onset, total wake time, sleep efficiency). Sleep efficiency was also obtained from wrist actigraphy. Subjective sleep quality was measured by the Pittsburgh Sleep Quality Index. Insomnia severity, depression and self-reported quality of life were measured as secondary outcomes. Data were analyzed for all randomized participants (n=159) in an intention to treat analysis. The study was not designed to compare differences in primary outcomes between individual and group CBT-I. Subjects who received individual and group CBT-I were pooled to form the intervention group. We hypothesized that the intervention would improve sleep (both objectively and subjectively) at six-month follow-up and improvements would be maintained at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Report symptoms that meet diagnostic criteria for insomnia and are:

* age >=60,
* community-dwelling,
* live within a 30-mile radius of VA Greater Los Angeles Healthcare System (GLAHS), and
* have transportation to VA GLAHS to attend the intervention/control programs.

Exclusion Criteria:

* Significant cognitive impairment (MMSE score <24) and have evidence of sleep apnea (by questionnaire and/or sleep monitoring).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy A. Alessi, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

REFERENCES:
- [Result] Fung CH, Martin JL, Igodan U, Jouldjian S, Alessi C. The association between difficulty using positive airway pressure equipment and adherence to therapy: a pilot study. Sleep Breath. 2013 May;17(2):853-9. doi: 10.1007/s11325-012-0779-y. Epub 2012 Nov 13. PMID 23149875
- [Result] Alessi C, Martin JL, Fiorentino L, Fung CH, Dzierzewski JM, Rodriguez Tapia JC, Song Y, Josephson K, Jouldjian S, Mitchell MN. Cognitive Behavioral Therapy for Insomnia in Older Veterans Using Nonclinician Sleep Coaches: Randomized Controlled Trial. J Am Geriatr Soc. 2016 Sep;64(9):1830-8. doi: 10.1111/jgs.14304. Epub 2016 Aug 22. PMID 27550552
- [Result] Fung CH, Martin JL, Josephson K, Fiorentino L, Dzierzewski JM, Jouldjian S, Song Y, Rodriguez Tapia JC, Mitchell MN, Alessi CA. Cognitive Expectancies for Hypnotic Use among Older Adult Veterans with Chronic Insomnia. Clin Gerontol. 2018 Mar-Apr;41(2):130-135. doi: 10.1080/07317115.2017.1356895. Epub 2017 Sep 29. PMID 28960164
- [Result] Hughes JM, Song Y, Fung CH, Dzierzewski JM, Mitchell MN, Jouldjian S, Josephson KR, Alessi CA, Martin JL. Measuring Sleep in Vulnerable Older Adults: A Comparison of Subjective and Objective Sleep Measures. Clin Gerontol. 2018 Mar-Apr;41(2):145-157. doi: 10.1080/07317115.2017.1408734. Epub 2017 Dec 28. PMID 29283797
- [Result] Yeung T, Martin JL, Fung CH, Fiorentino L, Dzierzewski JM, Rodriguez Tapia JC, Song Y, Josephson K, Jouldjian S, Mitchell MN, Alessi C. Sleep Outcomes With Cognitive Behavioral Therapy for Insomnia Are Similar Between Older Adults With Low vs. High Self-Reported Physical Activity. Front Aging Neurosci. 2018 Sep 13;10:274. doi: 10.3389/fnagi.2018.00274. eCollection 2018. PMID 30271340
- [Derived] Song Y, Kelly MR, Fung CH, Dzierzewski JM, Grinberg AM, Mitchell MN, Josephson K, Martin JL, Alessi CA. Change in Dysfunctional Sleep-Related Beliefs is Associated with Changes in Sleep and Other Health Outcomes Among Older Veterans With Insomnia: Findings From a Randomized Controlled Trial. Ann Behav Med. 2022 Jan 1;56(1):35-49. doi: 10.1093/abm/kaab030. PMID 33944909
- [Derived] Dzierzewski JM, Martin JL, Fung CH, Song Y, Fiorentino L, Jouldjian S, Rodriguez JC, Mitchell M, Josephson K, Alessi CA. CBT for late-life insomnia and the accuracy of sleep and wake perceptions: Results from a randomized-controlled trial. J Sleep Res. 2019 Aug;28(4):e12809. doi: 10.1111/jsr.12809. Epub 2019 Jan 4. PMID 30609099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from among community-dwelling older veterans who responded to an insomnia screening postal survey and who met diagnostic criteria for insomnia. The recruitment period was from May 2010 to February 2012. A total of 519 subjects were enrolled.
Pre-assignment Details: Following enrollment, subjects with a Mini-Mental State Exam (MMSE) score < 24 or an apnea hypopnea index (AHI) > 20 were ineligible for randomization. Subjects with unstable medical or psychological conditions were also excluded. Results are presented for the 159 subjects who were randomized (106 intervention and 53 control).
Groups:
- CBT-I: Manual-based cognitive behavioral therapy for insomnia (CBT-I) provided in 5 individual or group sessions by a health educator
Period: Overall Study
Arm/Group | CBT-I | Control
Started | 106 | 53
Completed | 89 | 51
Not Completed | 17 | 2
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Refused follow-up | 9 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who received individual and group intervention CBT-I were pooled to form the CBT-I intervention group.
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I | Control | Total
Number analyzed (Participants) | 106 | 53 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (7.9) | 72.4 (7.3) | 72.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 101 | 52 | 153

OUTCOME MEASURES:

1. Primary Outcome: Sleep Onset Latency
Description: Mean time to fall asleep based on 7-day sleep diary.
Time Frame: Six months after randomization
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | CBT-I | Control
Number analyzed (Participants) | 106 | 53
Minutes | 21.3 [16.8 to 25.8] | 31.3 [25.4 to 37.2]
Statistical Analysis 1: Comparison: CBT-I vs Control; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -15.8, 95% CI 2-sided [-28.7 to -3.0], Standard Error of Mean 6.6 — The parameter estimate is the improvement in sleep onset latency from baseline to 6-month follow-up for CBT-I group versus the same improvement in the control group

2. Primary Outcome: Wake After Sleep Onset
Description: Mean total minutes awake during nighttime awakenings based on 7-day sleep diary.
Time Frame: Six months after randomization
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | CBT-I | Control
Number analyzed (Participants) | 106 | 53
Minutes | 30.3 [22.9 to 37.7] | 42.8 [33.0 to 52.7]
Statistical Analysis 1: Comparison: CBT-I vs Control; Test type: Superiority; p = 0.21, Mixed Models Analysis; Mean Difference (Final Values) = -10.2, 95% CI 2-sided [-26.3 to 5.9], Standard Error of Mean 8.2 — The parameter estimate is the improvement in wake after sleep onset from baseline to 6-month follow-up for CBT-I group versus the same improvement in the control group

3. Primary Outcome: Total Wake Time
Description: Mean total minutes awake from bedtime to rise time based on 7-day sleep diary.
Time Frame: Six months after randomization
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | CBT-I | Control
Number analyzed (Participants) | 106 | 53
Minutes | 73.4 [61.4 to 85.4] | 108 [91.8 to 124.1]
Statistical Analysis 1: Comparison: CBT-I vs Control; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -37.0, 95% CI 2-sided [-62.2 to -11.7], Standard Error of Mean 12.9 — The parameter estimate is the improvement in total wake time from baseline to 6-month follow-up for CBT-I group versus the same improvement in the control group

4. Primary Outcome: Sleep Efficiency From Sleep Diary
Description: Sleep efficiency (mean percent time asleep while in bed) based on 7-day sleep diary.
Time Frame: Six months after randomization
Measure: Mean (95% Confidence Interval); unit: percentage of time asleep while in bed
Arm/Group | CBT-I | Control
Number analyzed (Participants) | 106 | 53
percentage of time asleep while in bed | 82.7 [81.3 to 84.1] | 83.1 [81.2 to 85.0]
Statistical Analysis 1: Comparison: CBT-I vs Control; Test type: Superiority; p = .005, Mixed Models Analysis; Mean Difference (Final Values) = 6.7, 95% CI 2-sided [2.0 to 11.3], Standard Error of Mean 2.36 — The parameter estimate is the improvement in sleep efficiency from baseline to 6-month follow-up for CBT-I group versus the same improvement in the control group

5. Primary Outcome: Sleep Efficiency From Wrist Actigraphy
Description: Sleep efficiency (mean percent time asleep while in bed) based on 7 days of wrist actigraphy.
Time Frame: Six months from randomization
Measure: Mean (95% Confidence Interval); unit: percentage of time asleep while in bed
Arm/Group | CBT-I | Control
Number analyzed (Participants) | 106 | 53
percentage of time asleep while in bed | 82.7 [81.3 to 84.1] | 83.1 [81.2 to 85.0]
Statistical Analysis 1: Comparison: CBT-I vs Control; Test type: Superiority; p = 0.15, Mixed Models Analysis; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-3.3 to 0.5], Standard Error of Mean 0.97 — The parameter estimate is the improvement in sleep efficiency (from wrist actigraphy) from baseline to 6-month follow-up for CBT-I group versus the same improvement in the control group

6. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index assesses subjective sleep quality and sleep disturbances The PSQI ia an 18-item questionnaire with a total score range from 0 - 21. A total score > 8 indicates poor sleep quality.
Time Frame: Six months after randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBT-I | Control
Number analyzed (Participants) | 106 | 53
units on a scale | 6.0 [5.3 to 6.7] | 7.2 [6.2 to 8.2]
Statistical Analysis 1: Comparison: CBT-I vs Control; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-3.5 to -1.3], Standard Error of Mean 0.55 — The parameter estimate is the improvement in PSQI score from baseline to 6-month follow-up for CBT-I group versus the same improvement in the control group

ADVERSE EVENTS:
Time Frame: From randomization to 12-month follow-up.
Arm/Group | CBT-I | Control
All-Cause Mortality (participants affected / at risk) | 3/106 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/53
Other Adverse Events (participants affected / at risk) | 0/106 | 0/53

LIMITATIONS AND CAVEATS:
The study sample was predominantly older male veterans, so results may not be generalizable to older women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No